CLINICAL TRIAL: NCT03744078
Title: A Randomized Trial of Foley Bulb and PGE2 for Labor Induction in Premature Rupture of Membranes
Brief Title: A Randomized Trial of Induction Methods in Premature Rupture of Membranes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Ahmet Eser, M.D., Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 47
Record Dates: First submitted 2018-03-27; First posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Preterm Premature Rupture of Fetal Membranes; Induction of Labor Affected Fetus / Newborn
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PGE2 with Foley balloon catheter (Active Comparator): 10 mg PGE2 vaginal ovul will be inserted to the posterior fornix and an 18-F Foley catheter which filling with 60 mL of saline solution will be placed into the cervix
  Interventions: Device: Foley balloon catheter
- PGE2 vaginal ovule (No Intervention): 10 mg PGE2 vaginal ovule will be inserted to the posterior fornix

INTERVENTIONS:
Device: Foley balloon catheter — 18-F Foley catheter which filling with 60 mL of saline solution will be placed into the cervix
  Arms: PGE2 with Foley balloon catheter

SUMMARY:
This study evaluates the addition of transcervical Foley catheter balloon and vaginal prostaglandin E2 induction in premature rupture of membranes. Half of participants will be used combine transcervical Foley catheter balloon and vaginal prostaglandin E2, while the other half will be used alone vaginal prostaglandin E2.

ELIGIBILITY:
Inclusion Criteria:

1. singleton pregnancy,
2. gestational age ≥34 weeks,
3. rupture of membranes,
4. cephalic presentation,
5. bishop score ≤5,
6. had less than three uterine contractions in every 10 minutes.

Exclusion Criteria:

1. Patients who had contraindications for vaginal delivery,
2. previous uterine surgery,
3. fetal malpresentation,
4. multifetal pregnancy,
5. more than three contractions in 10 minutes,
6. contraindications to prostaglandins,
7. a category II or III fetal heart rate pattern,
8. anomalous fetus,
9. fetal demise
10. women with immediate delivery indications -

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 200 (Estimated)
Dates: Start 2018-04-15 (Actual); Primary Completion 2018-12-15 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
induction-to- delivery time | an average of one year
  the length of time between the beginning of induction and the end of labor

SECONDARY OUTCOMES:
tachysystole | an average of one year
  uterine contractions more than 3 in 10 minutes
chorioamnionitis | an average of one year
  clinical chorioamnionitis(Maternal fever and Fetal tachycardia >160/min and Maternal tachycardia >100/min
postpartum hemorrhage | an average of one year
  abnormal uterine bleeding after birth
neonatal outcome | an average of one year
  APGAR scores
admission to neonatal intensive care unit | an average of one year
  admission to neonatal intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: ahmet eser, Study Director — Zeynep Kamil Maternity and Children's Training and Research Hospital, Department of Obstetrics and Gynecology, Istanbul, Turkey
Locations (2):
- Turkey (Türkiye) (2):
  - Doga, Istanbul, Kucukcekmece
  - Zeynep Kamil Education and Research Hospital, Istanbul, Uskudar

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264